CLINICAL TRIAL: NCT00795418
Title: A 52-week,Multi-center,Randomized,Double-blind,Placebo-controlled,Parallel Group Study in Patients With Mild Alzheimer's Disease to Investigate the Safety and Tolerability of Repeated Subcutaneous Injections of CAD106
Brief Title: Safety and Tolerability of Repeated Subcutaneous Injections of CAD 106 in Mild Alzheimer's Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCAD106A2202
Record Dates: First submitted 2008-11-10; First posted 2008-11-21 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2012-05

CONDITIONS: Alzheimer's Disease
Keywords: Active immunization; Alzheimer's disease; Antibody; Vaccine; Central Nervous System Diseases; Neurodegenerative diseases
MeSH Terms: conditions — Alzheimer Disease; Central Nervous System Diseases; Neurodegenerative Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- CAD106 (Experimental)
  Interventions: Biological: CAD106
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Placebo — Placebo comparator
  Arms: Placebo
Biological: CAD106
  Arms: CAD106

SUMMARY:
This study will evaluate the safety and tolerability of repeated subcutaneous injections of CAD106 in patients with mid Alzheimer's disease

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female patients between 40 and 85 years of age (both inclusive)
* Diagnosis of mild Alzheimer's Disease (AD)
* Mini-Mental State Examination (MMSE) 20 to 26 at screening, untreated or on stable dose of cholinesterase inhibitor or memantine over the last 6 weeks.

Exclusion Criteria:

* Previously participated in an AD vaccine study and received active treatment.
* History or presence of an active autoimmune and/or with an acute or chronic inflammation, and/or clinically relevant atopic condition.
* History or presence of seizures and/or cerebrovascular disease.
* Presence of other neurodegenerative disease and/or psychiatric disorders (with the exception of successfully treated depression)
* Advanced, severe, progressive or unstable disease that might interfere with the safety of the patient.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-10; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability of repeated injection of CAD106 at multiple timepoints including but not limited to screening, baseline and through the end of the study (adverse events, physical/neurologic exams, vital signs, 12- lead ECGs, clinical labs, brain MRI) | 52 weeks

SECONDARY OUTCOMES:
Immune response at multiple timepoints including but not limited to screening, baseline and through the end of the study. | 52 weeks
Cognitive assessments at multiple timepoints including but not limited to screening, baseline and through the end of the study. | 52 weeks
Functional assessments at multiple timepoints including but not limited to screening, baseline and through the end of the study. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- United States (10):
  - ATP Clinical Research, Costa Mesa, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Sunrise Clinical Research, Hollywood, Florida
  - Alexian Brothers Neuroscience Institute, Elk Grove Village, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - MidAmerica NeuroScience Research Foundation, Lenexa, Kansas
  - Columbia University Medical Center, New York, New York
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - NOCCR Knoxville, Knoxville, Tennessee
  - University of Texas Southwestern, Dallas, Texas

REFERENCES:
- [Derived] Farlow MR, Andreasen N, Riviere ME, Vostiar I, Vitaliti A, Sovago J, Caputo A, Winblad B, Graf A. Long-term treatment with active Abeta immunotherapy with CAD106 in mild Alzheimer's disease. Alzheimers Res Ther. 2015 Apr 27;7(1):23. doi: 10.1186/s13195-015-0108-3. eCollection 2015. PMID 25918556
- See also: Results for CCAD106A2202 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4704